CLINICAL TRIAL: NCT00395330
Title: Airways Dysfunction Following WTC Dust Exposure
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Other Study IDs: H06-714
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Diseases
Keywords: Respiratory Function Tests; Oscillometry; World Trade Center Disaster; Environmental Exposure; Distal Airways
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

SUMMARY:
In the weeks following the terrorist attacks of September 11, 2001, many patients presented to their physicians with complaints related to exposure to the debris. These included nose and throat complaints (drip, congestion, sore throat), increased GE reflux (heartburn, regurgitation, retrosternal chest burning) and respiratory symptoms (worsening cough, wheezing, shortness of breath, chest tightness, sleep disturbance). In addition, there was a disproportionate rate of self-reported worsening asthma symptoms in patients living in Lower New York 5-9 weeks after the attack; those with exposure to the dust cloud fared worse. The functional abnormalities of firefighters with exposures to dust at the WTC site has been recently described. However, the effects of WTC dust exposure on pulmonary function in residents and workers near the WTC site remain unclear. This study will retrospectively review the charts of all patients referred to the pulmonary function laboratory for evaluation of symptoms following exposure to WTC dust. The main objectives for this study will be to characterize the functional abnormalities in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80
* referral for pulmonary function evaluation of respiratory symptoms following exposure to WTC dust

Exclusion Criteria:

* inability to perform testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study will retrospectively review the charts of all patients referred to the pulmonary function laboratory for evaluation of symptoms following exposure to WTC dust.
Sampling Method: Non-Probability Sample
Enrollment: 500
Dates: Start 2003-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Berger, MD, Principal Investigator — NYU Langone Health

REFERENCES:
- [Derived] Oppenheimer BW, Goldring RM, Herberg ME, Hofer IS, Reyfman PA, Liautaud S, Rom WN, Reibman J, Berger KI. Distal airway function in symptomatic subjects with normal spirometry following World Trade Center dust exposure. Chest. 2007 Oct;132(4):1275-82. doi: 10.1378/chest.07-0913. Epub 2007 Sep 21. PMID 17890470